CLINICAL TRIAL: NCT01070537
Title: INVIBO: Evaluation of the Feasibility and Tolerance of an Intubation Procedure Performed by Means of the Bonfils Fiberscope in Awake Patients With Predicted Difficult Intubation in the Context of ENT Cancer Surgery
Brief Title: Evaluation of the Bonfils Fiberscope for Predicted Difficult Intubation in Awake Patients With Ear, Nose, and Throat (ENT) Cancer (INVIBO)
Acronym: INVIBO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Jean-Edgard MAZERES, Centre Léon Bérard - 28 rue Laennec - 69373 LYON Cedex 08 - France
Allocation: Not Applicable | Model: Single Group
Other Study IDs: INVIBO; ET2007-036 (Registry Identifier: CENTRE LEON BERARD)
Record Dates: First submitted 2010-02-15; First posted 2010-02-18 (Estimated); Last update posted 2010-02-18 (Estimated); Status verified 2010-02

CONDITIONS: Carcinoma
Keywords: Otolaryngology; Equipment and Supplies; Intubation
MeSH Terms: conditions — Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Bonfils fiberscope intubation

SUMMARY:
The Bonfils intubation fiberscope (BF), a rigid medical device with a curved tip, is exclusively used in anesthesiology for orotracheal intubation (OTI). The objective of the study was to evaluate the feasibility and the tolerance of an intubation procedure realized by means of the BF (BFI) in awake adult patients with predicted difficult intubation (PDI), in the context of ENT cancer surgery.

The intubation is performed under local anesthesia (either nasal, oral, or intercricothyroidal) and sedation using Remifentanyl (AIVOC) with spontaneous ventilation. The primary endpoint is the rate of BFI meeting quality requirements: the procedure must be both successful (≤ 2 attempts and duration < 180 sec) and well tolerated (Fahey score < 2). The secondary endpoints include the difficulties met by the operator during the BFI and patient's perception of the intubation procedure, evaluated in the recovery room and 7 days after the intervention. Sample size is calculated using a one-stage Fleming design with p0=80%, p1=95%, alpha=5% and 80% power, for a total of 32 evaluable patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged ≥ 18 years
* Requiring a surgical intervention for an ENT carcinoma
* Presenting with a PDI defined either as an Arne Score > 11, or a previous history of DI or by the surgeon's judgment.
* Able to understand, read and write French
* Signed, written informed consent

Exclusion Criteria:

* Impossible mask ventilation
* Patient with a laryngeal stridor indicative of upper airway stenosis
* Patient requiring an intubation by nasal route
* Glasgow score < 12
* BMI > 35
* Pregnant or lactating women
* Documented history of cognitive or psychiatric disorders
* Difficult follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2008-02; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
The rate of BFI meeting quality requirements: the procedure must be successful on the one hand (≤ 2 attempts and duration < 180 sec); and well tolerated on the other hand (Fahey score < 2). | 180 sec after the beginning of the intubation

SECONDARY OUTCOMES:
Number of well-tolerated BFI procedures | At the end of the intubation
Duration of the intubation procedure among patients with a successful BFI (≤ 2 attempts and duration < 180 sec) | At the end of the intubation
Frequency and type of difficulties met by the operator | At the end of the intubation
Frequency and type of adverse events experienced by the patient | At the end of the intubation
Patient's perception of the intubation procedure | In the recovery room and 7 days after the intubation

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Edgard Mazères, MD, Principal Investigator — Centre Leon Berard
Locations (1):
- Centre Léon Bérard, Lyon, France

REFERENCES:
- [Background] Benumof JL. Management of the difficult adult airway. With special emphasis on awake tracheal intubation. Anesthesiology. 1991 Dec;75(6):1087-110. doi: 10.1097/00000542-199112000-00021. PMID 1824555
- [Background] Arne J, Descoins P, Fusciardi J, Ingrand P, Ferrier B, Boudigues D, Aries J. Preoperative assessment for difficult intubation in general and ENT surgery: predictive value of a clinical multivariate risk index. Br J Anaesth. 1998 Feb;80(2):140-6. doi: 10.1093/bja/80.2.140. PMID 9602574
- [Background] Boisson-Bertrand D, Bourgain JL, Camboulives J, Crinquette V, Cros AM, Dubreuil M, Eurin B, Haberer JP, Pottecher T, Thorin D, Ravussin P, Riou B. [Difficult intubation. French Society of Anesthesia and Intensive Care. A collective expertise]. Ann Fr Anesth Reanim. 1996;15(2):207-14. No abstract available. French. PMID 8734245
- [Background] Halligan M, Charters P. A clinical evaluation of the Bonfils Intubation Fibrescope. Anaesthesia. 2003 Nov;58(11):1087-91. doi: 10.1046/j.1365-2044.2003.03407.x. PMID 14616594
- [Background] Bein B, Worthmann F, Scholz J, Brinkmann F, Tonner PH, Steinfath M, Dorges V. A comparison of the intubating laryngeal mask airway and the Bonfils intubation fibrescope in patients with predicted difficult airways. Anaesthesia. 2004 Jul;59(7):668-74. doi: 10.1111/j.1365-2044.2004.03778.x. PMID 15200542
- [Background] Bein B, Yan M, Tonner PH, Scholz J, Steinfath M, Dorges V. Tracheal intubation using the Bonfils intubation fibrescope after failed direct laryngoscopy. Anaesthesia. 2004 Dec;59(12):1207-9. doi: 10.1111/j.1365-2044.2004.03967.x. PMID 15549980
- [Background] Fahey MR, Morris RB, Miller RD, Sohn YJ, Cronnelly R, Gencarelli P. Clinical pharmacology of ORG NC45 (NorcuronTM): a new nondepolarizing muscle relaxant. Anesthesiology. 1981 Jul;55(1):6-11. doi: 10.1097/00000542-198107000-00003. PMID 6113794
- [Background] Cormack RS, Lehane J. Difficult tracheal intubation in obstetrics. Anaesthesia. 1984 Nov;39(11):1105-11. PMID 6507827
- [Background] Fleming TR. One-sample multiple testing procedure for phase II clinical trials. Biometrics. 1982 Mar;38(1):143-51. PMID 7082756
- [Background] Ramsay MA, Savege TM, Simpson BR, Goodwin R. Controlled sedation with alphaxalone-alphadolone. Br Med J. 1974 Jun 22;2(5920):656-9. doi: 10.1136/bmj.2.5920.656. PMID 4835444
- [Background] Mallampati SR, Gatt SP, Gugino LD, Desai SP, Waraksa B, Freiberger D, Liu PL. A clinical sign to predict difficult tracheal intubation: a prospective study. Can Anaesth Soc J. 1985 Jul;32(4):429-34. doi: 10.1007/BF03011357. PMID 4027773
- [Background] Loh KS, Irish JC. Traumatic complications of intubation and other airway management procedures. Anesthesiol Clin North Am. 2002 Dec;20(4):953-69. doi: 10.1016/s0889-8537(02)00022-6. PMID 12512271
- [Derived] Mazeres JE, Lefranc A, Cropet C, Steghens A, Bachmann P, Perol O, Rosay H. Evaluation of the Bonfils intubating fibrescope for predicted difficult intubation in awake patients with ear, nose and throat cancer. Eur J Anaesthesiol. 2011 Sep;28(9):646-50. doi: 10.1097/EJA.0b013e3283495b85. PMID 21743336